## **COVER PAGE**

| Official title of the study: | Laser acupuncture combined with |
|---|---|
| | acupressure improves low back pain and |
| | quality of life: a randomized controlled trial |
| NCT number: | No |
| Document date: | 26/04/2020 |

## Abstract

Background: Low back pain (LBP) is a common, huge health and socioeconomic health problem that affects physiological functions and reduces work efficiency in nurses.

Objective: This study aimed to evaluate the effect of low-level laser acupuncture combined with acupressure (LAA) on pain intensity, pain interference and life dysfunction in hospital nurses with LBP.

Methods: This single-blinded randomized controlled trial enrolled a convenience sample of nurses from one teaching hospital. Seventy-six participants were randomly assigned to the LAA group (n=38) receiving low-level laser acupuncture and auricular acupressure for four weeks, and a control group (n=38) receiving a similar intervention but without laser energy and acupressure. Data were collected using the Short Form of the Brief Pain Inventory (BPI-SF) and Roland-Morris Disability Questionnaire (RDQ) at three time points: baseline before the intervention, and Week 2 and Week 4 during the intervention.

Results: After controlling for prior low back pain, the result of linear mixed-effects model analysis showed trends in significant between-group differences, including: in worst pain occurring in Week 2 (p<0.001) and Week 4 (p<0.001); in current pain in Week 4 (p<0.001); in least pain in Week 2 (p=0.032) and Week 4 ( $\beta$ =-1.55, p<0.001); in pain interference in Week 2 (p=-0.009) and Week 4 (p<0.001); and in life dysfunction in Week 2 (p<0.001) and Week 4 ( $\beta$ =-3.95, p<0.001).

Conclusions: This study supports that the 4-week LAA intervention improves pain intensity, pain interference, and life dysfunction for hospital nurses with LBP. These effects were maintained continuously for at least 4 weeks after the intervention. The LAA may be another effective, easy-to-use, non-invasive nonpharmacological

analgesic intervention for low back pain.



Flow chart of research design and participant allocation

BPI-SF: Short Form of the Brief Pain Inventory, RMDQ: Roland Morris Disability Questionnaire.

(This article under submission)